CLINICAL TRIAL: NCT05497466
Title: PUMCH Study Into Individualized Scanning for Coronary Artery Disease
Acronym: COE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-2806 COE V1.3
Record Dates: First submitted 2022-07-31; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease; Coronary Computed Tomographic Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects who are male or female outpatients aged 18 years and scheduled for CCTA to rule out CAD: 300 patients scheduled for coronary CTA examination to rule out CAD in PUMCH. Each subject will be selected and assigned in a specific tube-voltage arm by the scanner based on the patient's body habitus for individualized CTA scans, without any intervention

SUMMARY:
Cardiac computed tomographic angiography (CCTA) is a non-invasive diagnostic imaging technique for visualization of the coronary arteries and thus, frequently used in the evaluation of coronary artery disease (CAD). CT technology is improving continuously, and various technological advances not only increase diagnostic accuracy, but also provide a substantial reduction in radiation dose and scan acquisition time. These modifications challenge optimal synchronization and timing of scan protocols in CM administration due to a shorter data acquisition window, hereby creating opportunities for injection strategies with a decrease in total amount of contrast media (CM). [4-6] Reducing the radiation dose of CT angiography and injected CM dose have become a routine need and trend in clinical practice. In addition to this, physical factors such as cardiac output and body weight are considered important factors with regard to variability in vascular enhancement. A standard 'one size fits all' protocol with a standard injected CM volume, independent of weight and length of the patient has proven to be outdated and precision medicine in the future should be based on individually tailored scan and CM injection protocols that are more scientific and involve various parameters such as individual tube voltage, patients weight and heart rate to benefit patients by reducing radiation exposure and CM dose while fulfilling the diagnostic purpose.

Prospective studies focused on modifying both scan and injection parameters were completed in the Dutch (representing European) patient population with body weight varying between 40 and 130kg by Maastricht University Medical Center (MUMC) and have shown very promising results in Dutch population. In theory, these scan and injection protocols should be applicable to both average Dutch population (e.g. European population) and other heterogeneous patient populations, i.e. world-wide patient populations with any BMI category. However, so far, the effectiveness of this approach has not been deliberately discussed in the (on average) heavier North American population or the lighter Asian population. So, prior to promotion of the individually tailored CT scan protocols for global use, we need to obtain enough evidence in terms of the diagnostic confidence from those protocols in Chinese patients who could represent Asian population.

DETAILED DESCRIPTION:
Primary objective: To prospectively evaluate the diagnostic quality (including the intravascular attenuation of the coronary arteries and image quality) in a previously validated individualized scan and CM injection CCTA protocol whereas both scan and injection parameters are tailored to the individual patient in Chinese population.

Secondary Objective(s):

1. To evaluate the radiation dose and contrast media dose of this individualized approach for CCTA in a Chinese patient population.
2. To evaluate the injection parameters required for the average patient population.

Subjects will be screened according to clinical data and enrolled in the study after providing informed consent. Patients will be scanned by Siemens Force CT scanner, prospective ECG gate-control and narrow window scanning technology, as well as intelligent KV (CARE-KV Tech) scanning technology. The CARE-kV software will determine optimal scan parameters for each patient, without any human intervention. By this means, each patient will be included in a specific tube-voltage arm based on in the condition of individual patient.

Care kV is a software that collects information about the patient's own attenuation values/ x-ray absorption during a so-called scout scan. Based on these parameters and taking into account the required scan quality (e.g. parenchymal, bone or vascular), the software determines the optimal scan settings for the patient. This includes both a variable tube current (in mAs) along the z-axis of the patient and an individual tube voltage (in kV). The tube voltage can be selected between 70 and 150kV in steps of 10kV. For this study, the scan quality slider will be set to 'vascular' or '11', which is commonly used in clinical studies and clinical practice for CCTA.

Iopromide injection (iodine concentration 370 mgI/ml) (Ultravist, Bayer Healthcare, Berlin, Germany) is administered as a bolus through the cubital vein using dual-syringe high-pressure injector (CT high-pressure injector: Stellant, MEDRAD, Pittsburg, PA, USA). The CM injection parameters are computed according to patient and examination-related parameters (patient weight, CM concentration, scan duration and maximum flow rate) using the Personalized Patients Protocol Technology (P3T) software supplied in the high-pressure injector.

P3T (Personalized Patient Protocol Technology) software computes individualized contrast injection protocols. P3T Cardiac/Pulmonary arteries are indicated for use with CAT of the cardiac structures, coronary arteries, chambers of the heart, pulmonary vasculature, thoracic and abdominal aorta. During initial setup, options such as minimum and maximum iodine loads, minimum injection duration, and other settings are configured according to site preferences and guidelines. These options are stored as a "preset", which can then be selected to calculate an injection protocol. At that time, patient and procedure specific parameters (patient weight, CM concentration, scan duration, and maximum flow rate) are entered by the radiographer. The software calculates the iodine load by multiplying the patient weight by a pre-determined dosing factor, applying the configured minimums and maximums. Then, the injection duration is determined based on the duration of the scan and minimum injection duration. Using the iodine load, injection duration, and CM concentration, the individualized flow rate and CM volumes are computed. The radiographer may edit the injection protocol if necessary. Dosing factors were derived based on pharmacokinetic model to simulate vascular enhancement in the regions of interest, targeting 350-400 HU across a wide range of patients.

An 18G or 20G venous access in the antecubital vein is preferred for higher flow rates. If low flow rates are required, venous access through an IV needle as small as 22G (max flow: 6.5 mL/sec) may be used.

* Test bolus + saline flush, next CM bolus and saline flush 40ml. Prewarmed (37 º C [99˚F]) CM (Iopromide 370mgI/ml, Bayer).
* Injection using a programmable dual-head CT injector (Stellant, Bayer), via an 18-20G intravenous injection catheter in the left or right antecubital vein. We propose to use the appropriate gauge for the expected flow rate, according to local safety regulations.
* P3T Cardiac Certegra/ Use patient body weight adjusted protocol: P3T Cardiac, Certegra. (This will show flow rates if one sets the injection time and contrast media concentration).
* Adjust for selected kV setting by adapting the IDR: -10% for 110kV, -20% for 100kV, -30% for 90kV, -40% for 80kV and -50% for 70kV.
* In all patients, a test bolus injection at the level of the ascending aorta is performed to assess optimal start delay; 20ml of CM at a flow rate according to P3T protocol. Test bolus is followed by 40ml of saline flush at the same flow rate.

Study archiving: patient protocol (radiation dose information), ECG information, contrast media information, scout views calcium score scan, heart scan (Bv40, 0.6mm slices).

For this study we chose to include 300 patients to ensure a representation of normal patient variance. Given the assumed non-diagnostic rate to be around 5%, the 95% CI of non-diagnostic rate with 300 sample size is [2.8 %, 8.1%]. Although there is no hypothesis test planned for this study, the result from a recent published study taking similar design on individualized scan and injection protocol of liver CT provides support on adequate sample size of the current study. Based on the study, 256 patients in total could enable the stratification performed based on age (<60 and ≥60 years) and weight (<75 and ≥75 kg) in the population weighed below 115 kg.

If 300 patients are not included after 18 months, the inclusion period will be over none the less.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patient aged older than 18;
* Deny previous cardiovascular history；
* Atypical or typical complaints of angina and referred for CCTA to rule out CAD with Iopromide 370 mgI/ml by clinicians
* Possibility of 'flash' mode scan: patient heart rate below 70 beats per minute and regular rhythm；
* Patients or families are able to understand the study protocol and willing to participate in the study and provide written informed consent.

Exclusion Criteria:

* Any contraindications for prospective ECG gate-control CT coronary angiography, including：

  1. Inability to perform a breath hold for at least the expected scan time；
  2. Unstable angina；
  3. Hemodynamic instability；
  4. Pregnant or lactating women；
  5. Renal insufficiency (defined as eGFR<30 ml/min/1.73m2);
  6. Previous history of adverse reactions to iodinated contrast agents；
  7. Confirmed or suspected hyperthyroidism or pheochromocytoma；
  8. Atrial fibrillation or arrhythmia; severe congestive heart failure (class IV according to NYHA classification of cardiac function)；
* History of CAD
* Patients undergoing PCI before coronary CTA examination, or patients with a previous history of heart bypass surgery
* Insufficient cannula venous access (preferred 18G, minimal 20G cannula)；
* Patients who are participating other clinical studies。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to consecutively include 300 patients scheduled for coronary CTA examination to rule out CAD in PUMCH.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic quality produced by individualized scan and injection protocol. | 48 hours post examination
  When using an individualized scan and injection protocol, definition of diagnostic quality of the scan is the imaging result could satisfy the following two criteria：
  1. Intravascular attenuation of the target coronary arteries should be over 325 Hounsfield Units (HU).
  2. Subjective overall image quality should be diagnostic (image quality > 2 of a 5-point Likert scale).

SECONDARY OUTCOMES:
Objective evaluation on image quality | 48 hours post examination
  The images are transferred to the Siemens image processing workstation for post-processing. The post-vascular enhancement CT value of chambers of the heart, aorta and all branch vessels of coronary arteries is measured with standard deviation (SD) as image noise; the CT value of the inferior wall myocardium is measured with SD as background noise. Signal-To-Noise Ratio (SNR) is calculated as follows: SNR=enhanced CT value/SD.
Subjective evaluation on image quality | 48 hours post examination
  According to the 17-segment coronary artery segmentation standards of the American Heart Association, the images are scored by two radiologists who are blinded to protocol and have more than 5 years of work experience in CCTA with the 5-point Likert scale for scoring of coronary artery image quality: 5 points (excellent), images have fine anatomical details, sharp edges, and no obvious noise; 4 points (good), images have fine anatomical details and slightly increased noise; 3 points (fair), the visualization of most of anatomical results on the image satisfies diagnostic needs, with obvious but acceptable noise; 2 points (poor), images have blurred anatomical details that are difficult to distinguish and obvious noise; 1 point (very poor), images have extremely obvious noise that results in failed diagnosis.
contrast media dose in ml | During Injection procedure
  injection parameters will be continuously monitored and automatically measured by a data acquisition program, Certegra™ Informatics Platform (Bayer Healthcare, Berlin, Germany). The contrast media dose could be recorded and read out directly in the system.
contrast media flow rate in ml/s | During Injection procedure
  injection parameters will be continuously monitored and automatically measured by a data acquisition program, Certegra™ Informatics Platform (Bayer Healthcare, Berlin, Germany). Contrast media flow rate could be recorded and read out from the system.
contrast media peak flow rate [ml/s] | During Injection procedure
  injection parameters will be continuously monitored and automatically measured by a data acquisition program, Certegra™ Informatics Platform (Bayer Healthcare, Berlin, Germany). The peak flow rate could be recorded and read out from the system
Time-to-peak of contrast media [s] | During Injection procedure
  injection parameters will be continuously monitored and automatically measured by a data acquisition program, Certegra™ Informatics Platform (Bayer Healthcare, Berlin, Germany). Time to peak of contrast media could be recorded and read out from the system
iodine delivery rate (IDR) in mgI/s | During Injection procedure
  IDR= concentration of contrast media (mgI/ml) administrated X flow rate(ml/s).injection parameters will be continuously monitored and automatically measured by a data acquisition program, Certegra™ Informatics Platform (Bayer Healthcare, Berlin, Germany). IDR of contrast media could be read out from the system.
Patient radiation dose:volume CT dose index (CTDIvol) in mGy | 48 hours post examination
  Radiation parameters will be continuously monitored and automatically measured by a data acquisition programs Radimetrics Enterpise Platforms (Bayer Healthineers, Berlin, Germany). CTDIvol could be read out directly from the system.
Patient radiation dose: size-specific dose estimates (SSDEs) of chest in mGy | 48 hours post examination
  Radiation parameters will be continuously monitored and automatically measured by a data acquisition programs Radimetrics Enterpise Platforms (Bayer Healthineers, Berlin, Germany). SSDEs of chest could be read out directly from the system
Patient radiation dose: dose length product (DLP) in mGy*cm | 48 hours post examination
  Radiation parameters will be continuously monitored and automatically measured by a data acquisition programs Radimetrics Enterpise Platforms (Bayer Healthineers, Berlin, Germany). DLP could be read out from the system.
Patient radiation dose: effective dose (ED) in mSv | 48 hours post examination
  Radiation parameters will be continuously monitored and automatically measured by a data acquisition programs Radimetrics Enterpise Platforms (Bayer Healthineers, Berlin, Germany). ED could be read out from the system.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengyu Jin, Principal Investigator — PUMCH

IPD SHARING:
Plan to Share IPD: Undecided
There is a rule in China, for sharing any individual patient information, the study responsible must get authority's approval